CLINICAL TRIAL: NCT01341769
Title: A Study to Determine the Effects of Added Ingredients on Glycaemic and Insulinemic Responses to a Snack Food
Brief Title: Blood Glucose and Insulin Responses to Snack Food Products
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Test ingredient production did not meet specification
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Reading Scientific Services Ltd. (Industry)
Responsible Party: Richard Black, Ph.D., VP, Nutrition and Peter H. Brown, Ph.D., Research Principal, Nutrition Research, Kraft Foods, Inc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P10-08857 version 01
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Study Focus 1:Glycaemic Index; Study Focus 2:Glycaemic Response; Study Focus 3:Insulinemic Response
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Test Food (Placebo Comparator): Snack base
  Interventions: Other: Dietary Intervention
- Experimental Test Food 1 (Experimental): Snack Base containing ingredient 1
  Interventions: Other: Dietary Intervention
- Experimental Test Food 2 (Experimental): Snack base containing ingredient 2
  Interventions: Other: Dietary Intervention
- Experimental Test Food 3 (Experimental): Snack base containing ingredients 1 and 2
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention
  Arms: Control Test Food
Other: Dietary Intervention
  Arms: Experimental Test Food 1
Other: Dietary Intervention
  Arms: Experimental Test Food 2
Other: Dietary Intervention
  Arms: Experimental Test Food 3

SUMMARY:
The purpose of this study is to assess the effects of added food ingredients, when baked into a snack food product, on glycaemic index of the product and glycaemic and insulinemic responses to the product in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not less than 40% males or females
* Non-smoker
* Aged 18 to 55 years
* Have a body mass index between 18.5 to 29.99 kg/m2
* Fasting blood glucose (finger-stick) >3.3 and <5.6 mmol/L (Visit 2)
* Two-hour OGTT glucose (finger-stick) <7.8 mmol/L (Visit 2)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Females who are lactating or may be pregnant or if of childbearing potential, are not taking adequate contraceptive precautions
* Any significant concurrent illness
* History of allergy likely to interfere with the study or known sensitivity to the test food or its ingredients
* Have assessed an investigational product for GI in the last 72 hours.
* Concurrent participation in any other safety study
* History of diabetes, hepatitis, AIDS, anaemia or a heart condition
* The use of any medication or dietary supplement which might, in the opinion of the principal investigator 1) make participation in the study dangerous to the subject, or 2) may affect the results.
* Had any type of gastrointestinal surgery, including gastric bypass
* Having consumed anything apart from plain water in the 12 hours prior to each test
* Have been medically diagnosed as having high blood pressure or heart disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Glycaemic index of experimental test foods compared to that of control test food using venous plasma. | 0-120 minutes

SECONDARY OUTCOMES:
Glycaemic index of experimental test foods compared to that of control test food using capillary blood | 0-120 minutes
Determine and compare glycaemic responses to experimental test foods and control test food using venous plasma and capillary blood | 0-180 minutes
Measure insulin in venous plasma | 0-180 minutes
Measure C-peptide in venous plasma | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Hart, SCS, Dip, MICR, Study Director — Reading Scientific Services Limited; Dr. Suzana Louth, Principal Investigator — Reading Scientific Services Limited
Locations (1):
- Reading Scientific Services Limited, Reading, Berkshire, United Kingdom